CLINICAL TRIAL: NCT07402499
Title: Validity and Reliability of an Immersive Virtual Reality Adaptation of the Timed Up and Go Test in Individuals With Chronic Non-Specific Low Back Pain
Brief Title: Validation of a Virtual Reality Timed Up and Go Test in Adults With Chronic Non-Specific Low Back Pain
Acronym: VRTUG-CLBP
Status: Not yet recruiting | Type: Observational
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Mehmet Akif Guler, Lecturer Dr., Selcuk University
Other Study IDs: SU-SBF-FTR-VRTUG-2026-001
Record Dates: First submitted 2026-02-04; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Chronic Low Back Pain
Keywords: Virtual Reality; Timed Up and Go Test; Functional Mobility; Validity; Reliability; Test-Retest; Oswestry Disability Index; Pain Measurement; Kinesiophobia; Tampa Scale for Kinesiophobia
MeSH Terms: conditions — Kinesiophobia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chronic Non-Specific Low Back Pain Group: Adults aged 18-55 years with chronic non-specific low back pain who undergo functional mobility assessment using the Timed Up and Go test and its virtual reality adaptation (VR-TUG).

SUMMARY:
This study evaluates whether an immersive virtual reality (VR) version of the Timed Up and Go (TUG) test can accurately measure functional mobility in adults with chronic non-specific low back pain.

The standard TUG test measures the time needed to stand up from a chair, walk 3 meters, turn around, walk back, and sit down. In the VR version (VR-TUG), participants perform the same movements while wearing a VR headset that displays a virtual environment.

We will examine: (1) whether VR-TUG results are similar to the standard TUG, (2) whether VR-TUG is reliable when repeated about one week later, and (3) whether VR-TUG performance is associated with pain, disability, and fear of movement.

Participants will complete questionnaires (VAS, ODI, and TSK), perform standard TUG and VR-TUG at baseline, and repeat VR-TUG 7 ± 2 days later. Results will help determine whether VR-based functional mobility testing is a practical assessment tool for people with chronic low back pain.

DETAILED DESCRIPTION:
BACKGROUND:

Chronic non-specific low back pain (CNSLBP) is a leading cause of disability worldwide. The Timed Up and Go (TUG) test is a valid and reliable measure of functional mobility in individuals with musculoskeletal conditions, including chronic low back pain, and TUG performance has been shown to correlate with pain intensity and disability. Virtual reality (VR) has increasingly been used as a therapeutic intervention for chronic low back pain, but the use of immersive VR as an assessment tool has not been systematically evaluated in this population.

STUDY DESIGN:

This is a prospective, single-center, observational methodological study designed to assess the validity and test-retest reliability of an immersive virtual reality adaptation of the Timed Up and Go test (VR-TUG) in individuals aged 18-55 years with chronic non-specific low back pain.

PROCEDURES:

* Session 1 (Baseline Assessment):

  * Demographic and clinical data collection
  * Pain intensity (Visual Analog Scale, VAS)
  * Functional disability (Oswestry Disability Index, ODI - validated Turkish version)
  * Kinesiophobia (Tampa Scale for Kinesiophobia - Turkish version)
  * Classic TUG test performance
  * VR-TUG test performance (first measurement)
* Session 2 (7 ± 2 days later):

  * VR-TUG test performance (second measurement for test-retest reliability)

VR-TUG PROTOCOL:

Participants will wear a head-mounted display (HMD) that presents an immersive virtual environment replicating the spatial parameters of the classic TUG test. They will perform the same sequence of movements (stand up from a chair, walk 3 meters forward, turn 180°, walk back, and sit down) while immersed in the virtual environment. Time to completion will be recorded. A brief familiarization period (approximately 1-2 minutes) will be provided before testing. Participants will be monitored for any adverse effects (such as dizziness, nausea, or visual discomfort), and the VR-TUG will be stopped immediately if needed.

OUTCOME MEASURES:

* Primary Outcome:

  o VR-TUG completion time (seconds), including assessment of test-retest reliability across two sessions.
* Secondary Outcomes:

  * Classic TUG completion time (seconds)
  * Pain intensity (VAS)
  * Functional disability (ODI)
  * Kinesiophobia (Tampa Scale for Kinesiophobia)

ANALYSIS PLAN:

* Concurrent validity:

  o Correlation between VR-TUG and classic TUG completion times (Pearson or Spearman correlation, depending on data distribution).
* Test-retest reliability:

  * Intraclass correlation coefficient (ICC, two-way mixed-effects model, single measure) for VR-TUG completion time between Session 1 and Session 2.
  * Estimation of standard error of measurement (SEM) and minimal detectable change (MDC).
  * Bland-Altman analysis to evaluate agreement between repeated VR-TUG measurements.
* Construct validity:

  * Correlations between VR-TUG completion time and clinical measures (VAS, ODI, Tampa Scale for Kinesiophobia). It is expected that longer VR-TUG times will be associated with higher pain, disability, and kinesiophobia scores.

Statistical significance will be set at p < 0.05.

SAMPLE SIZE:

Based on previous studies reporting excellent reliability of technology-supported functional tests in patients with chronic low back pain (ICC ≥ 0.90), a sample size of approximately 65 participants was calculated to detect a correlation of 0.70 between classic TUG and VR-TUG with 90% power and an alpha of 0.05, allowing for potential dropouts.

SAFETY CONSIDERATIONS:

All testing will be conducted in a safe, obstacle-free environment under the supervision of a trained researcher who can provide physical support if needed. Participants will be screened for contraindications to VR use (for example, photosensitive epilepsy or severe motion sickness). Testing will be stopped immediately if participants experience significant discomfort, dizziness, increased pain, loss of balance, or any other adverse effect. All adverse events and reasons for test discontinuation will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 55 years.
* Clinician-diagnosed chronic non-specific low back pain (pain duration ≥ 3 months).
* Applied to Selcuk University Medical Faculty Physical Therapy and Rehabilitation outpatient clinic with low back pain complaint.
* Able to walk independently and safely perform the Timed Up and Go (TUG) and VR-TUG tests (with or without usual assistive device).
* Able to understand and follow instructions; literate in Turkish (at least primary school education).
* Willing to participate and able to provide written informed consent.

Exclusion Criteria:

* Red flag conditions or suspected specific pathology (e.g., fracture, tumor/metastasis, infection such as spondylitis/discitis).
* Inflammatory back pain suggestive of conditions such as ankylosing spondylitis or sacroiliitis.
* Significant radiculopathy or neurological deficit (dermatomal leg pain, marked weakness, reflex changes, sensory loss), clinically significant lumbar disc herniation, severe spinal stenosis, or spondylolisthesis grade II or higher.
* Prior lumbar spine surgery.
* Lower-extremity conditions that substantially limit mobility (e.g., severe hip/knee osteoarthritis, hip/knee arthroplasty, amputation, severe deformity).
* Neurological disorders affecting gait or balance (e.g., stroke, Parkinson's disease, multiple sclerosis, progressive neuromuscular disease).
* Vestibular disorder or recurrent severe vertigo affecting balance.
* Severe cardiac or pulmonary disease that may compromise safety during testing.
* Pregnancy.
* Contraindications to VR use (e.g., photosensitive epilepsy) or history of severe VR intolerance (significant nausea, dizziness, visual discomfort, or migraine triggered by VR).
* Severe cognitive impairment, major psychiatric disorder, or communication problems preventing cooperation.
* Severe visual or hearing impairment that prevents following instructions or safely using VR.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Adults aged 18-55 years with clinician-diagnosed chronic non-specific low back pain who present to the Selcuk University Medical Faculty Physical Therapy and Rehabilitation outpatient clinic and meet the eligibility criteria.
Sampling Method: Probability Sample
Enrollment: 65 (Estimated)
Dates: Start 2026-03-21 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Virtual Reality Timed Up and Go (VR-TUG) Completion Time | Baseline and 7 ± 2 days (test-retest)
  Time (in seconds) to complete the VR-adapted Timed Up and Go test while wearing a head-mounted display, including standing from a chair, walking 3 meters, turning 180°, walking back, and sitting down.

SECONDARY OUTCOMES:
Timed Up and Go (TUG) Completion Time | Baseline
  Time (in seconds) to complete the standard Timed Up and Go test.
Pain Intensity (Visual Analog Scale, VAS) | Baseline
  Pain intensity measured using a 10-cm visual analog scale (score 0-10).
Disability (Oswestry Disability Index, ODI) | Baseline
  Self-reported disability related to low back pain measured with the Oswestry Disability Index (ODI), Turkish validated version (score 0-100).
Kinesiophobia (Tampa Scale for Kinesiophobia, TSK) | Baseline
  Fear of movement/(re)injury measured with the Tampa Scale for Kinesiophobia (TSK), Turkish version (score 17-68).

OTHER OUTCOMES:
Test-Retest Reliability of VR-TUG (ICC) | Baseline and 7 ± 2 days
  Intraclass correlation coefficient (two-way mixed-effects, single measure) for VR-TUG completion time between baseline and 7 ± 2 days.
Agreement and Measurement Error of VR-TUG (SEM/MDC, Bland-Altman) | Baseline and 7 ± 2 days
  Standard error of measurement (SEM), minimal detectable change (MDC), and Bland-Altman agreement analyses for VR-TUG completion time across two sessions.

CONTACTS AND LOCATIONS:
Locations (1):
- Selcuk University Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Konya, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) that underlie the primary and secondary outcome results of this study will be shared. This includes the analyzable dataset containing demographic variables, VR-TUG and TUG completion times, pain intensity (VAS), disability (ODI), kinesiophobia scores, and key covariates used in the main analyses.
Supporting Information: Study Protocol, SAP
Time Frame: De-identified IPD and supporting documents will be available after publication of the primary outcome results and will remain available for 3 years thereafter.
Access Criteria: De-identified IPD will be made available to qualified researchers upon reasonable request. Requests must include a methodologically sound proposal and will be reviewed by the study team. Data sharing will comply with institutional and ethical guidelines, and a data use agreement may be required.

REFERENCES:
- [Background] Tunca, Ö. Y., Yakut, Y., Uygur, F., & Uluğ, N. (2011). Tampa Kinezyofobi Ölçeği'nin Türkçe versiyonu ve test-tekrar test güvenirliği. Fizyoterapi Rehabilitasyon, 22(1), 44-49.
- [Background] Yakut E, Duger T, Oksuz C, Yorukan S, Ureten K, Turan D, Frat T, Kiraz S, Krd N, Kayhan H, Yakut Y, Guler C. Validation of the Turkish version of the Oswestry Disability Index for patients with low back pain. Spine (Phila Pa 1976). 2004 Mar 1;29(5):581-5; discussion 585. doi: 10.1097/01.brs.0000113869.13209.03. PMID 15129077
- [Background] Ozsoy G, Aksoy K. Intra- and inter- rater reliability of the face-to-face assessment and tele-assessment of performance-based tests in older adults. Eur Geriatr Med. 2024 Jun;15(3):601-607. doi: 10.1007/s41999-024-00946-7. Epub 2024 Feb 21. PMID 38383819
- [Background] Delbes L, Mascret N, Goulon C, Montagne G. Validation of an immersive virtual reality device accepted by seniors that preserves the adaptive behavior produced in the real world. Front Bioeng Biotechnol. 2022 Sep 2;10:917486. doi: 10.3389/fbioe.2022.917486. eCollection 2022. PMID 36118569
- [Background] Muhla F, Clanche F, Duclos K, Meyer P, Maiaux S, Colnat-Coulbois S, Gauchard GC. Impact of using immersive virtual reality over time and steps in the Timed Up and Go test in elderly people. PLoS One. 2020 Mar 13;15(3):e0229594. doi: 10.1371/journal.pone.0229594. eCollection 2020. PMID 32168361
- [Background] Garay-Sanchez A, Suarez-Serrano C, Ferrando-Margeli M, Jimenez-Rejano JJ, Marcen-Roman Y. Effects of Immersive and Non-Immersive Virtual Reality on the Static and Dynamic Balance of Stroke Patients: A Systematic Review and Meta-Analysis. J Clin Med. 2021 Sep 28;10(19):4473. doi: 10.3390/jcm10194473. PMID 34640491
- [Background] Huang G, Chen W. Therapeutic effects of virtual reality technology on chronic low back pain. Medicine (Baltimore). 2025 Nov 7;104(45):e45867. doi: 10.1097/MD.0000000000045867. PMID 41204536
- [Background] Hirano K, Imagama S, Hasegawa Y, Ito Z, Muramoto A, Ishiguro N. Impact of low back pain, knee pain, and timed up-and-go test on quality of life in community-living people. J Orthop Sci. 2014 Jan;19(1):164-71. doi: 10.1007/s00776-013-0476-0. Epub 2013 Oct 17. PMID 24132792
- [Background] Moreno-Ligero M, Duenas M, Failde I, Del Pino R, Coronilla MC, Moral-Munoz JA. Psychometric Properties of the Pictorial Pain Interference Questionnaire for Assessing Functional Interference in Chronic Low Back Pain. Arch Phys Med Rehabil. 2024 Oct;105(10):1870-1879. doi: 10.1016/j.apmr.2024.05.029. Epub 2024 Jun 10. PMID 38866224
- [Background] Buraschi R, Pollet J, Villafane JH, Piovanelli B, Negrini S. Temporal and kinematic analyses of timed up and go test in chronic low back pain patients. Gait Posture. 2022 Jul;96:137-142. doi: 10.1016/j.gaitpost.2022.05.027. Epub 2022 May 26. PMID 35635989
- [Background] Dobson F. Timed Up and Go test in musculoskeletal conditions. J Physiother. 2015 Jan;61(1):47. doi: 10.1016/j.jphys.2014.11.003. Epub 2014 Dec 10. No abstract available. PMID 25497269
- [Background] Podsiadlo D, Richardson S. The timed "Up & Go": a test of basic functional mobility for frail elderly persons. J Am Geriatr Soc. 1991 Feb;39(2):142-8. doi: 10.1111/j.1532-5415.1991.tb01616.x. PMID 1991946
- [Background] Maher C, Underwood M, Buchbinder R. Non-specific low back pain. Lancet. 2017 Feb 18;389(10070):736-747. doi: 10.1016/S0140-6736(16)30970-9. Epub 2016 Oct 11. PMID 27745712
- [Background] Vlaeyen JWS, Maher CG, Wiech K, Van Zundert J, Meloto CB, Diatchenko L, Battie MC, Goossens M, Koes B, Linton SJ. Low back pain. Nat Rev Dis Primers. 2018 Dec 13;4(1):52. doi: 10.1038/s41572-018-0052-1. PMID 30546064